CLINICAL TRIAL: NCT03067675
Title: Topcon DRI OCT Triton Reference Database Study
Brief Title: Triton Reference Database
Status: Completed | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Triton RDB
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Healthy Eyes
Keywords: no known ocular pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects Presenting With Normal Eyes: Subjects with no known ocular diseases will be scanned on the Topcon DRI OCT Triton (plus) device
  Interventions: Device: Topcon DRI OCT Triton (plus)

INTERVENTIONS:
Device: Topcon DRI OCT Triton (plus) — OCT Machine used for diagnostic purposes

SUMMARY:
The objective of this study is to collect OCT measurement data on normal healthy eyes.

DETAILED DESCRIPTION:
The objective of this study is to collect OCT measurement data on normal healthy eyes in order to determine the reference limits for Topcon DRI OCT Triton based on the percentile points for 1%, 5%, 95%, and 99%.

ELIGIBILITY:
Inclusion Criteria

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with normal eyes bilaterally (cataracts are acceptable)
4. IOP ≤ 21 mmHg bilaterally
5. BCVA 20/40 or better bilaterally

Exclusion Criteria

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images
3. HFA visual field (24-2 Sita Standard, white on white) result unreliable (based on manufacturer's recommendation), defined as fixation losses > 20% or false positives > 33%, or false negatives > 33%
4. Visual field defects consistent with glaucomatous optic nerve damage based on at least one of the following two findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   2. Glaucoma hemi-field test "outside normal limits."
5. Narrow angle
6. History of leukemia, dementia or multiple sclerosis
7. Concomitant use of hydroxychloroquine and chloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of subjects without eye disease.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Retinal Thickness | 1 Minute
  The thickness of the macula layer

CONTACTS AND LOCATIONS:
Overall Officials: Charles Riesman, MS, Study Chair — Topcon Corporation
Locations (6):
- United States (6):
  - Southern California College of Optometry, Anaheim, California
  - Accessoreyes Optometry, Pasadena, California
  - Illinois College of Optometry, Chicago, Illinois
  - Fischer Laser Eye Center, Willmar, Minnesota
  - New York VA, Jamaica, New York
  - Stat University of New York College of Optometry, New York, New York

IPD SHARING:
Plan to Share IPD: No